CLINICAL TRIAL: NCT01664585
Title: EXERCISE TRAINING WITH PHYSICALLY ACTIVE LIFESTYLE TO REDUCE HEADACHE AND INCREASE QUALITY OF LIFE. A Randomised Controlled Trial of the Effectiveness and Cost-effectiveness of Exercise Training and Physical Activity on Chronic Headache
Brief Title: Exercise Training With Physically Active Lifestyle to Reduce Headache and Quality of Life
Acronym: HEADEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Jyväskylä Central Hospital (Other); University of Jyvaskyla (Other)
Responsible Party: Principal Investigator, Marjo Rinne, PhD, Researcher, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R12006; UKK Institute/173 (Other Grant/Funding Number: Kela-The Social Insurance Institution of Finland/36/26/2011)
Record Dates: First submitted 2012-08-07; First posted 2012-08-14 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Headache; Physical Activity; Quality of Life
Keywords: headache; women; exercise; fear avoidance; physical activity
MeSH Terms: conditions — Headache; Motor Activity | interventions — Sensitivity Training Groups; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (Experimental): The rationale and means for the exercise program are to
  1. Motivate and teach participants for postural and motor control and strengthening exercises
  2. Monitor and motivate to continue exercise training, and to increase their physical activity
  Training is organised six times as a 60-min session during six months: two individually supervised sessions, and four following training sessions will be accomplished in groups of 10 participants guided by an experienced physical therapist. Three weekly similar home training sessions are recommended for participants. Information on amount of exercise sessions per week and repetitions of each exercise will be collected via exercise diary. To perform home training, a DVD and/or booklet will be provided to participants in the training group.
  Interventions: Behavioral: Training group
- Control (Sham Comparator): The control group will receive six sessions of Transcutaneous Nervous Stimulation treatment (TNS) as a placebo treatment (0), and the participants in this group are recommended and encouraged to maintain their previous normal level of physical activity and exercise habits throughout the study without any supervision or home training programs.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Training group — The 60-minute training sessions include a few mobilization techniques for upper neck. In detail, three different exercises concentrated on postural and motor control will be taught during the first two training sessions. Progressively, two additional exercise movements aiming at postural and motor control will be taught in the next session. After eight weeks, two muscle strength exercises utilising therapeutic rubber band will be included into the program. The aim of the rubber band exercises is eventually to achieve the load of 80% of maximal voluntary contraction. The participants in the training group are also instructed to increase their amount of physical activity progressively according to the current physical activity recommendations.
  Other Names: Movement control of neck; Muscle training of the postural muscles of upper neck; Physical activity
  Arms: Training group
Behavioral: Control — The control group will receive six sessions of Transcutaneous Nervous Stimulation treatment (TNS) as a placebo treatment (0) and the participants in control group are recommended and encouraged to maintain their previous normal level of physical activity and exercise habits throughout the study without any supervision or home training programs.
  Arms: Control

SUMMARY:
The aim of this intervention study is to examine whether tailored exercise therapy training is effective and cost-effective to decrease headache frequency and intensity, reduce medication used for chronic headache and patients´ absence from work, improve their neck muscle force, cervical spine mobility, functional ability and quality of life, and increase general physical activity in chronic headache women at regular work during a 6-month intervention.

The intervention itself with pilot-tested upper-neck specific exercise regimen aims that patients would independently commit to train and exercise to reduce their headache, and thus increase their quality of life. In addition, reduced pain and frequency of headache may increase the objectively measured daily physical activity of chronic headache patients.

DETAILED DESCRIPTION:
Tension-type,migraine and cervicogenic headache are the most common reasons for visits to a primary care physician among working women. Headache has major economic impact due to patients' absence from work, and pharmacy claims. Neck symptoms induce three percent of all visits to a primary care physician and 1 % of all costs in health care, and moreover, institutionalizing increase costs of treatment. Active treatment may offer cost-effective option for outpatients. In addition, there is no data showing how much headache/neck pain restricts participation in physical activity (PA) or other activities in society.

The purpose of this study is to investigate whether specific therapeutic exercises reduce cervicogenic headache cost-effectively, and simultaneously improve neck function and quality of life. The other aim is to evaluate the effect of exercises on daily PA in women with chronic headache.

The following hypotheses will be tested:

1. Specific therapeutic exercises based on individual training reduce cost-effectively cervicogenic headache and improve neck function, and quality of life on women at regular work during a 6-month intervention
2. The intervention increases general physical activity of women with cervicogenic headache
3. The intervention assists them to manage the headache by way of exercising during the follow-up.
4. Physical activity of women with chronic cervicogenic headache is lower than average in Finnish population.

The HEADEX intervention study is a randomized controlled trial. Volunteers, women at regular work and having ongoing status with chronic migraine and/or cervicogenic headache will be recruited using newspaper advertising, from the register of Finnish Migraine Society and occupational health care services in Helsinki, Tampere and Jyvaskyla. The study sample is restricted to women, as the headache is much more common in women. After recruitment, the eligibility of patients to participate is screened. In total, the aim is to obtain 120 women to participate. The two subsequent baseline assessments and follow-up of headaches with the diary between two months before the beginning of the intervention enable ensuring intensity and type of the headache and that it is chronic. Randomisation is centralised but the intervention will be accomplished and clustered in three study centres. Sample size has been estimated for the primary outcomes. The number of participant will be 60 women in treatment and 60 control group.

The 6 months exercise intervention consists of 6 supervised progressive exercise training sessions and home training program, and the participants are instructed to increase their PA. The main emphasis of the exercise program is to improve and relearn postural and movement control of neck, and later on strengthen the postural muscles. The exercise intervention consists of six supervised progressive exercise training sessions to teach rehabilitative training technique with similar home training program. Before the intervention, information on work ergonomics will be enquired and if needed, changes will be recommended. The control group will receive Transcutaneous Nervous Stimulation treatment (6 times) as a placebo treatment (intensity 0), and recommendation to maintain their PA at previous level. The follow-up is identical for both groups, and information on exercise frequency is collected up to 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 to 60 and currently at work and aim to continue at same work at least two years
* intensity of headache on Visual Analog Scale (VAS) has been equal or greater than 45 mm (scale 0-100) during last two months
* Headache Impact Test TM [HIT-6 Scoring Interpretation Finland (Finnish) Version 1.1] 58/78 points

Exclusion Criteria:

* severe degenerative changes at cervical vertebra or discus (including discus prolapse)
* whiplash injury or injury, which is contraindication for exercise and active lifestyle
* treated with manual therapy or physiotherapy within a previous month
* changed medication known to affect headaches during a previous month
* changed bifocals during previous month
* athletic trainees (3 or more times per week)
* alcoholic and/or drug addicts/ AUDIT The Alcohol Use Disorders Identification Test, Finnish version
* mental depression

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2015-07-03 (Actual); Study Completion 2015-07-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in headache intensity at 6 months | At baseline and follow-up after 6-months intervention
  The intensity of pain caused by headache is measured with Visual Analogue Scale (VAS)which is a measurement instrument for subjective experience. The participants specify their level of pain by indicating a position along a continuous line between two end-points (0 to 100).

SECONDARY OUTCOMES:
Amount and intensity of weekly physical activity | At baseline, after 6-mo, 12-mo,and 24-mo
  Objective assessment of daily physical activity during 7 days by accelerometer
Health economics | At baseline, after 6-mo, 12-mo, and 24-mo
  To evaluate the cost-effectiveness the calculations will be based on the self-reported absence from work (off work because of headache, possible disability pension because of headache), cost of medical and pharmaceutical claims for headache, ergonomic changes at work ergonomic changes at work, and adverse events of training. Furthermore, the costs of the intervention including the salaries of the study personnel, individual grants for the members of the research team, and costs related to examination of the subjects are entered to the total costs.
Quality of Life (QoL) | At baseline, after 6-mo, 12-mo, and 24-mo
  The data will be collected with RAND-36 quality of life questionnaires , the FACT Fatigue scale and mood, and the Beck depression inventory (BDI).
Fear avoidance beliefs | At baseline, after 6-mo, 12-mo, and 24-mo
  Changes in fear-avoidance behaviour will be assessed with questionnaire on fear-avoidance beliefs (FABQ) addressing the behaviour both in work and leisure (Waddell et. al 1993)
Frequency of headache | At baseline, after 6-mo, 12-mo, and 24-mo
  Participants keep diaries on daily basis in terms of number of headache periods and mail the diaries to the investigator every month,
Disability | At baseline, after 6-mo, 12-mo, and 24-mo
  The participants will complete the Neck Disability Index (NDI)questionnaire with questions of ADL functioning

CONTACTS AND LOCATIONS:
Overall Officials: Marjo B Rinne, PhD, Study Director — UKK Institute; Riku P Nikander, PhD, Principal Investigator — University of Jyvaskyla; Arja H Häkkinen, PhD, Principal Investigator — University of Jyvaskyla; Jari J Ylinen, MD, DO, PhD, Principal Investigator — Jyväskylä Central Hospital; Katriina Kukkonen-Harjula, MD, Principal Investigator — Rehabilitation, South Karelia Social and Health Care District (Eksote); Kari Tokola, MSci, Principal Investigator — UKK Institute; Sanna Garam, MSci, Principal Investigator — Helsinki Metropolia University of Applied Sciences
Locations (3):
- Finland (3):
  - University of Jyväskylä, Jyväskylä
  - Jyväskylä Central Hospital, Department of Physical and Rehabilitation Medicine, Jyväskylä
  - UKK Institute, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Hertogh W, Vaes P, Devroey D, Louis P, Carpay H, Truijen S, Duquet W, Oostendorp R. Preliminary results, methodological considerations and recruitment difficulties of a randomised clinical trial comparing two treatment regimens for patients with headache and neck pain. BMC Musculoskelet Disord. 2009 Sep 23;10:115. doi: 10.1186/1471-2474-10-115. PMID 19775434
- [Background] Fricton J, Velly A, Ouyang W, Look JO. Does exercise therapy improve headache? a systematic review with meta-analysis. Curr Pain Headache Rep. 2009 Dec;13(6):413-9. doi: 10.1007/s11916-009-0081-2. No abstract available. PMID 19889280
- [Background] Fuller G, Kaye C. Headaches. BMJ. 2007 Feb 3;334(7587):254-6. doi: 10.1136/bmj.39090.652847.DE. No abstract available. PMID 17272568
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL. Manipulation or mobilisation for neck pain. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004249. doi: 10.1002/14651858.CD004249.pub3. PMID 20091561
- [Background] Jull G, Trott P, Potter H, Zito G, Niere K, Shirley D, Emberson J, Marschner I, Richardson C. A randomized controlled trial of exercise and manipulative therapy for cervicogenic headache. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1835-43; discussion 1843. doi: 10.1097/00007632-200209010-00004. PMID 12221344
- [Background] Ylinen J, Takala EP, Nykanen M, Hakkinen A, Malkia E, Pohjolainen T, Karppi SL, Kautiainen H, Airaksinen O. Active neck muscle training in the treatment of chronic neck pain in women: a randomized controlled trial. JAMA. 2003 May 21;289(19):2509-16. doi: 10.1001/jama.289.19.2509. PMID 12759322
- [Background] Ylinen J, Kautiainen H, Wiren K, Hakkinen A. Stretching exercises vs manual therapy in treatment of chronic neck pain: a randomized, controlled cross-over trial. J Rehabil Med. 2007 Mar;39(2):126-32. doi: 10.2340/16501977-0015. PMID 17351694
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Result] British Association for the Study of Headache Guidelines for All Healthcare Professionals in the Diagnosis and Management of Migraine, Tension-Type, Cluster and Medication-Overuse Headache Writing Committee: EA MacGregor, TJ Steiner, PTG Davies 3rd edition (1st revision). 2010.